CLINICAL TRIAL: NCT03239249
Title: Systematic Follow-up in Order to Reduce Drop-out in Upper Secondary Schools: A Cluster-randomized Evaluation of the IKO-model
Brief Title: The Cluster-randomized Evaluation of the IKO-model
Acronym: IKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian ministry of Education and Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48657 (NSD)
Record Dates: First submitted 2017-06-06; First posted 2017-08-04 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2020-09

CONDITIONS: School Drop Out Prevention
Keywords: school dropout prevention; intervention study; cluster-randomized
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Of all schools (42) in four counties, 20 have been randomized to experimental and 22 have been randomized to control condition. Schools randomized to experimental condition implement the IKO-model, while schools randomized to control condition work with drop-out as previously.
Who Masked: Participant
Masking Description: Students and guardians are masked for experimental condition, teachers and collaborating professionals are not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: IKO-model (20 schools) (Experimental): Schools randomized to experimental group will implement the IKO-drop-out prevention intervention. Each county have a project leader responsible for following up the implementation. The model is described in a manual, that schools should follow.
  Interventions: Other: IKO-model
- Treatment as usual (22 schools) (Active Comparator): Schools randomized to control group will work as previously with their drop-out prevention. This include various activities, but they are not systematic as in the IKO-model.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: IKO-model — A systematic model for drop-out prevention.
  Arms: Intervention group: IKO-model (20 schools)
Other: Treatment as usual — Schools randomized to control group (22) work as previously with school dropout
  Arms: Treatment as usual (22 schools)

SUMMARY:
The aim of this study is to analyze whether and how a systemic school-level approach to dropout prevention (the IKO-model), increase the completion rate from upper secondary school. The hypothesis is that schools that implement the model (i.e. randomized to the experimental group), will reduce the amount of students in risk of dropout, compared to their counterparts in schools randomized to the control group. The main expected outcomes in the study are; 1) increased amounts of students in upper secondary education completing their education within the three-year standard length of education, 2) decreased amounts of school-drop out, and 3) reduced values in mediating variables, such as low achievement, course failures, lack of attendance and lack of school-motivation and -effort. Accordingly, implementation quality and fidelity to the model will be assessed, both with quantitative (survey) and qualitative (interviews and observation) data. A total of five counties and 42 upper secondary schools participate in the evaluation project. One of the counties (Akershus County) have developed and piloted the model and function as a mentor in the other four counties (Oppland, Hedmark, Nord-Trøndelag and Hamar). While 20 schools have been randomized to the experimental group, 22 schools have been randomized to the control group. Schools randomized to the control group will work as earlier with school dropout.

DETAILED DESCRIPTION:
The aim of this study is to analyze whether and how a systemic school-level approach to dropout prevention (the IKO-model), increase the completion rate from upper secondary school. The hypothesis is that schools that implement the model (i.e. randomized to the experimental group), will reduce the amount of students in risk of dropout, compared to their counterparts in schools randomized to the control group. The main expected outcomes in the study are; 1) increased amounts of students in upper secondary education completing their education within the three-year standard length of education, 2) decreased amounts of school-drop out, and 3) reduced values in mediating variables, such as low achievement, course failures, lack of attendance and lack of school-motivation and -effort. Accordingly, implementation quality and fidelity to the model will be assessed, both with quantitative (survey) and qualitative (interviews and observation) data. A total of five counties and 42 upper secondary schools participate in the evaluation project. One of the counties (Akershus County) have developed and piloted the model and function as a mentor in the other four counties (Oppland, Hedmark, Nord-Trøndelag and Hamar). While 20 schools have been randomized to the experimental group, 22 schools have been randomized to the control group. Schools randomized to the control group will work as earlier with school dropout.

The implemented model is based on the County of Akershus´ experiences of developing and implementing the IKO-model since 2009. The IKO-model represents a systemic intervention at the school-level level, with the aim of improving the schools' follow-up structures related to students in risk of school dropout.

The basic idea of the model is that there are three groups of students: 1) students with ordinary follow-up needs, 2) students with the right to special education and 3) students without the right to special education, but who need individually targeted efforts from time to time. While there are guidelines and requirements when it comes to the follow-up of students with the right to special education, schools are less systematic in their approaches to students with temporary need for follow-up. Hence, the IKO-model focuses on improving the way schools identify and follow-up students in risk for dropout, but who do not qualify for special education. It is also emphasized, that time-limited and low-cost interventions are sufficient enough to reduce the risk of drop-out for the majority of students within this group, however the most important is to identify problems early and find solutions quickly. The goal is to remove the need for additional interventions as soon as possible and return students to normal education.

Another assumption is that the model will help schools to implement goal-focused targeted interventions at an early stage and ensure that the measures implemented are adjusted based on student needs. At student level the model aim to a) early identify students "in risk" for drop-out , b) charter students´ situation in order to find suitable interventions, and c) follow-up identified students with immediate interventions including an ongoing evaluation of their situation. In order for schools to succeed at identifying, chartering and following-up students, three main school-level components are implemented; 1) a computer assisted early warning system, 2) organizational structures and practices that enables schools to monitor progress and implement effective interventions, and 3) external and school internal communities of learning.

The research question is whether, how and to what extent the IKO-model reduce drop-out from upper secondary school. The hypothesis is that the IKO-model will assist schools in their work with identifying, charting and supporting students in risk through the early warning system, organization-level monitoring practices, and communities of learning. The main outcome assessed is reduced amounts of students that dropout from upper secondary school measured through increased amounts of students accomplishing education within the three-year standard length. The intervention is also expected to reduce amounts of students not in education, activity or employment at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 42 upper secondary schools in 4 Norwegian counties participate in the evaluation project.
* All first grade students in 2016 and 2017 arre followed up in the project.
* All first grade teachers are included in the study.

Exclusion Criteria:

NA

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7678 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the amount of students accomplishing their education within 3 years | 3 years after baseline measurement (T1)
  Administrative data delivered from the counties
change in the level of absence for students | baseline data (prior to randomization) compared to +12, +24 and +36 months after baseline
  Level of absence in upper secondary school, measured by administrative data
change in grades (maths, norwegian, english) | baseline data (prior to randomization) compared to +12, +24 and +36 months after baseline
  improved grades in upper secondary school, measured by administrative data

SECONDARY OUTCOMES:
change in school motivation | comparison between baseline data (T1) and follow-up 18 months later
  A Norwegian scale measuring school motivation
change in school achievement | comparison between baseline data (T1) and follow-up 18 months later
  Harters self-perception profile for adolescents

CONTACTS AND LOCATIONS:
Locations (42):
- Norway (42):
  - Arendal videregående skole, Arendal, Aust-Agder Fylkeskommune
  - Sam Eyde videregående skole, Arendal, Aust-Agder
  - Dahlske videregående skole, Grimstad, Aust-Agder
  - Setesdal videregående skole, Hornnes, Aust-Agder
  - Møglestu videregående skole, Lillesand, Aust-Agder
  - Risør videregående skole, Risør, Aust-Agder
  - Tvedestrand og Åmli videregående skole, Tvedestrand, Aust-Agder
  - Storsteigen videregående skole, Alvdal, Hedmark
  - Solør videregående skole, Braskereidfoss, Hedmark
  - Ringsaker videregående skole, Brumunddal, Hedmark
  - Elverum videregående skole, Elverum, Hedmark
  - Hamar katedralskole, Hamar, Hedmark
  - Storhamar videregående skole, Hamar, Hedmark
  - Midt-Østedal videregående skole, Koppang, Hedmark
  - Skarnes videregående skole, Skarnes, Hedmark
  - Jønsberg videregående skole, Stange, Hedmark
  - Stange videregående skole, Stange, Hedmark
  - Trysil videregående skole, Trysil, Hedmark
  - Nord-Østedal videregående skole, Tynset, Hedmark
  - Grong videregående skole, Grong, Nord-Trøndelag
  - Inderøy videregående skole, Inderøy, Nord-Trøndelag
  - Leksvik videregående skole, Leksvik, Nord-Trøndelag
  - Levanger videregående skole, Levanger, Nord-Trøndelag
  - Meråker videregående skole, Meråker, Nord-Trøndelag
  - Olav Duun videregående skole, Namsos, Nord-Trøndelag
  - Mære landbruksskole, Sparbu, Nord-Trøndelag
  - Steinkjer videregående skole, Steinkjer, Nord-Trøndelag
  - Ole Vig videregående skole, Stjørdal, Nord-Trøndelag
  - Verdal videregående skole, Verdal, Nord-Trøndelag
  - Dokka videregående skole, Dokka, Oppland
  - Gjøvik videregående skole, Gjøvik, Oppland
  - Hadeland videregående skole, Gran, Oppland
  - Nord Gulbrandsdalen videregående skole, Gulbrandsdalen, Oppland
  - Valdres videregående skole, Leira, Oppland
  - Lena-Valle videregående skole, Lena, Oppland
  - Lillehammer videregående skole, Lillehammer, Oppland
  - Raufoss videregående skole, Raufoss, Oppland
  - Vinstra videregående skole, Vinstra, Oppland
  - Gausdal videregående skole, Østre Gausdal, Oppland
  - Sentrum videregående skole, Kongsvinger
  - Øvrebyen videregående skole, Kongsvinger
  - Ytre Namdal videregående skole, Rørvik

IPD SHARING:
Plan to Share IPD: No